CLINICAL TRIAL: NCT02811276
Title: A Randomized, Controlled, Cross-over Trial Investigating the Impact of a High Protein Diet on Substrate Oxidation and Energy Metabolism in Healthy Women
Brief Title: The Impact of a High Protein Diet on Substrate Oxidation and Energy Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Almased Wellness GmbH (Industry)
Responsible Party: Principal Investigator, Carla Prado, Assistant Professor; CAIP Chair in Nutrition, Food and Health; and Director of the Human Nutrition Research Unit, University of Alberta
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00066006
Record Dates: First submitted 2016-06-16; First posted 2016-06-23 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Dietary Modification
Keywords: High-protein diet; Energy metabolism; Substrate oxidation
MeSH Terms: interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Those assigned to the Control Group will receive a eucaloric diet (a diet designed to meet the person's energy needs and maintain body weight) composed of 55% of carbohydrate, 15% of protein, and 30% of lipid.
- High-Protein Diet Group (Experimental): Those assigned to the High-Protein Diet Group will receive a eucaloric diet composed of 35% of carbohydrate, 40% of protein, and 25% of lipid constructed around a soy protein-based meal replacement (Almased®).
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — The High-Protein Diet Group will receive a eucaloric diet composed of 35% of carbohydrate, 40% of protein, and 25% of lipid constructed around a soy protein-based meal replacement (Almased®) for one and a half day. Participants will consume 1 gram ± 0.1 of Almased® per kg of body weight mixed with linseed oil and skim milk in their breakfast, lunch and dinner. Two snacks (afternoon and evening) composed of 1 gram ± 0.1 of Almased® per kg of body weight mixed with vegetable juice and linseed oil will also be provided.
  Arms: High-Protein Diet Group

SUMMARY:
In the 19th century, researchers found out that the differences in the energy content of macronutrients (protein, carbohydrate and fat) can elicit different responses in the amount of calories individuals burn per day. It was demonstrated that protein has a metabolic advantage when compared to the other macronutrients (carbohydrate and fat). Since these findings, researchers all over the world started to study how diets differing in macronutrient distribution could result in different responses to energy metabolism. Diets with high amounts of protein (i.e. meats, eggs, dairy products, and grains) are becoming more popular, and studies have shown that when people eat high quantities of protein they lose weight and fat mass, maintain the weight loss, and burn more calories per day.

The investigators hypothesize that giving high amounts of protein to healthy women will increase the amount of calories and fat they burn per day, increase their satiety, and improve health markers when compared to a normal diet. The increased protein level will be achieved using a nutrition supplement consisted of soy protein, yogurt and honey.

To test this, the investigators plan to divide the participants in two groups: one will eat a normal diet and the other a diet with high amounts of protein during one and a half day. After one month they will change groups and eat the other diet for the same period of time. During this period consuming the diets (1.5 days), participants will stay inside a whole body calorimetry suite, which is similar to a hotel bedroom and is able to inform in the most precise way the amount of calories participants will burn and if they are burning more fat. Additionally, before and after each meal participants will have to answer a questionnaire about their appetite sensations and blood will also be collected to analyze health markers.

DETAILED DESCRIPTION:
The aim of this study is to investigate the impact of a high protein diet (achieved through the use of a high protein supplement) versus standard diet on substrate oxidation and energy expenditure using a state-of-the-art live-in whole body calorimetry unit (WBCU).

This study will be an acute randomized, controlled, cross-over trial. Healthy women (n=24) will receive a run-in diet for three days and will then be randomly allocated into one of the following groups: 1) Control group receiving an eucaloric standard diet (55% of carbohydrate, 15% of protein, and 30% of lipid); 2) High-protein group: eucaloric high protein diet (35% of carbohydrate, 40% of protein, and 25% of fat) constructed around a soy protein-based meal replacement. The wash-out period will be of approximately one month. While receiving the diets in the WBCU for 32 hours, participants' overall change in energy metabolism including respiratory quotient will be assessed. Additional assessments include metabolic blood markers (glucose, insulin, lipid panel, peptide tyrosine-tyrosine, ghrelin, leptin, free glycerol, and free fatty acids), and appetite sensations (hunger and satiety). Body composition and energy requirements will be assessed at baseline using dual-energy X-ray absorptiometry and indirect calorimetry, respectively.

It is expected that the high-protein diet will increase lipid oxidation, and energy expenditure, with other favorable changes in the additional markers when compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy;
* Non-smoker;
* Female;
* Aged 18 to 34.9 years;
* Body mass index (BMI) between 18.5 and 24.9 kg/m² (preferably between 20 and 24.9 kg/m²);
* Regular menstrual cycle (lasting between 25 and 35 days).

Exclusion Criteria:

* Have previously been diagnosed with any kind of disease;
* Are taking any medications which may alter energy metabolism or body composition;
* Are lactose, gluten and/or soy allergic/intolerant;
* Follow a vegetarian, vegan or restrictive dietary pattern;
* Are pregnant or lactating;
* Have used nutritional supplements in the past two months;
* Perform over an hour per day of leisure time physical activity or more than seven hours per week of strenuous activity;
* Have had a nuclear medicine scan or injection of an X-ray dye in the past week;
* Have had a barium test/exam in the last two weeks;
* Claustrophobia.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Difference in fat balance assessed by indirect calorimetry during 32 hours of a high-protein (HP) total diet replacement compared to 32hours of a control (CON) diet. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  To measure the differences in fat balance during 32 hours of a high-protein (HP) total diet replacement compared to 32hours of a control (CON) diet.

SECONDARY OUTCOMES:
Difference in 24-hour energy expenditure assessed by indirect calorimetry during 32 hours of a high-protein (HP) total diet replacement compared to 32hours of a control (CON) diet. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  To measure the differences in 24-hour energy expenditure during 32 hours of a high-protein (HP) total diet replacement compared to 32 hours of a control (CON) diet.

OTHER OUTCOMES:
Changes in appetite sensations assessed by a 100 mm visual analogue scale questionnaire. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  Changes in hunger, satiety, fullness, and prospective food consumption will be rated by participants on a 100 mm visual analogue scale immediately before and 30 minutes after each meal and snack provided while participants spend 32 hours inside the whole body calorimetry unit while receiving a high-protein diet or a control diet. The 100 mm visual analogue scale is administered using the paper-and-pen method and participants are instructed to make a single vertical mark at the appropriate point between the two anchors on each scale to indicate the intensity of their subjective states regarding each element (between 0 and 100 mm):
  Hunger: 0 mm = "I am not hungry at all"; 100 mm = "I have never been more hungry".
  Satiety: 0 mm = "I am completely empty"; 100 mm = "I cannot eat another bite". Fullness: 0 mm = "Not at all full"; 100 mm = "Totally full". Prospective food consumption: 0 mm = "Nothing at all"; 100 mm = "A lot".
Changes in blood glucose levels. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  Changes in glucose will be assessed four times (fasting on the first day - at 07:45 a.m.; after the exercise session on the first day - at 11:00 a.m.; two hours postprandial on the first day - at 02:30 p.m.; fasting on the second day - at 08:30 a.m.) while participants spend 32 hours inside the whole body calorimetry unit while receiving a high-protein diet or a control diet.
Changes in blood insulin levels. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  Changes in insulin will be assessed four times (fasting on the first day - at 07:45 a.m.; after the exercise session on the first day - at 11:00 a.m.; two hours postprandial on the first day - at 02:30 p.m.; fasting on the second day - at 08:30 a.m.) while participants spend 32 hours inside the whole body calorimetry unit while receiving a high-protein diet or a control diet.
Changes in blood lipid panel levels. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  Changes in lipid panel will be assessed four times (fasting on the first day - at 07:45 a.m.; after the exercise session on the first day - at 11:00 a.m.; two hours postprandial on the first day - at 02:30 p.m.; fasting on the second day - at 08:30 a.m.) while participants spend 32 hours inside the whole body calorimetry unit while receiving a high-protein diet or a control diet.
Changes in blood peptide tyrosine-tyrosine levels. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  Changes in peptide tyrosine-tyrosine will be assessed four times (fasting on the first day - at 07:45 a.m.; after the exercise session on the first day - at 11:00 a.m.; two hours postprandial on the first day - at 02:30 p.m.; fasting on the second day - at 08:30 a.m.) while participants spend 32 hours inside the whole body calorimetry unit while receiving a high-protein diet or a control diet.
Changes in blood glucagon-like peptide-1 levels. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  Changes in glucagon-like peptide-1 will be assessed four times (fasting on the first day - at 07:45 a.m.; after the exercise session on the first day - at 11:00 a.m.; two hours postprandial on the first day - at 02:30 p.m.; fasting on the second day - at 08:30 a.m.) while participants spend 32 hours inside the whole body calorimetry unit while receiving a high-protein diet or a control diet.
Changes in blood ghrelin levels. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  Changes in ghrelin will be assessed four times (fasting on the first day - at 07:45 a.m.; after the exercise session on the first day - at 11:00 a.m.; two hours postprandial on the first day - at 02:30 p.m.; fasting on the second day - at 08:30 a.m.) while participants spend 32 hours inside the whole body calorimetry unit while receiving a high-protein diet or a control diet.
Changes in blood leptin levels. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  Changes in leptin will be assessed four times (fasting on the first day - at 07:45 a.m.; after the exercise session on the first day - at 11:00 a.m.; two hours postprandial on the first day - at 02:30 p.m.; fasting on the second day - at 08:30 a.m.) while participants spend 32 hours inside the whole body calorimetry unit while receiving a high-protein diet or a control diet.
Changes in blood free glycerol levels. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  Changes in glycerol will be assessed four times (fasting on the first day - at 07:45 a.m.; after the exercise session on the first day - at 11:00 a.m.; two hours postprandial on the first day - at 02:30 p.m.; fasting on the second day - at 08:30 a.m.) while participants spend 32 hours inside the whole body calorimetry unit while receiving a high-protein diet or a control diet.
Changes in blood free fatty acids levels. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  Changes in free fatty acids will be assessed four times (fasting on the first day - at 07:45 a.m.; after the exercise session on the first day - at 11:00 a.m.; two hours postprandial on the first day - at 02:30 p.m.; fasting on the second day - at 08:30 a.m.) while participants spend 32 hours inside the whole body calorimetry unit while receiving a high-protein diet or a control diet.
Difference in energy expenditure assessed by indirect calorimetry during 32 hours of a high-protein (HP) total diet replacement compared to 32hours of a control (CON) diet. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  To measure the differences in selected components of energy expenditure (resting, basal, sleep and postprandial - kcal) during 32 hours of a high-protein (HP) total diet replacement compared to 32 hours of a control (CON) diet.
Difference in substrate oxidation assessed by indirect calorimetry during 32 hours of a high-protein (HP) total diet replacement compared to 32hours of a control (CON) diet. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  To measure the differences in substrate oxidation rates (carbohydrate and protein - grams per day) during 32 hours of a high-protein (HP) total diet replacement compared to 32 hours of a control (CON) diet.
Difference in substrate balance assessed by indirect calorimetry during 32 hours of a high-protein (HP) total diet replacement compared to 32hours of a control (CON) diet. | During a 32-hour period while receiving a HP total diet replacement or a CON diet.
  To measure the differences in substrate balance (carbohydrate and protein - grams per day) during 32 hours of a high-protein (HP) total diet replacement compared to 32 hours of a control (CON) diet.

CONTACTS AND LOCATIONS:
Overall Officials: Carla MM Prado, PhD, Principal Investigator — University of Alberta; Arya Sharma, PhD, Principal Investigator — Unviersity of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oliveira CLP, Boule NG, Elliott SA, Sharma AM, Siervo M, Berg A, Ghosh S, Prado CM. A high-protein total diet replacement alters the regulation of food intake and energy homeostasis in healthy, normal-weight adults. Eur J Nutr. 2022 Jun;61(4):1849-1861. doi: 10.1007/s00394-021-02747-1. Epub 2021 Dec 20. PMID 34928408
- [Derived] Oliveira CLP, Boule NG, Sharma AM, Elliott SA, Siervo M, Ghosh S, Berg A, Prado CM. A high-protein total diet replacement increases energy expenditure and leads to negative fat balance in healthy, normal-weight adults. Am J Clin Nutr. 2021 Feb 2;113(2):476-487. doi: 10.1093/ajcn/nqaa283. PMID 33247306
- [Derived] Oliveira CLP, Boule NG, Sharma AM, Elliott S, Siervo M, Ghosh S, Berg A, Prado CM. Examining the effects of a high-protein total diet replacement on energy metabolism, metabolic blood markers, and appetite sensations in healthy adults: protocol for two complementary, randomized, controlled, crossover trials. Trials. 2019 Dec 27;20(1):787. doi: 10.1186/s13063-019-3950-y. PMID 31881910